CLINICAL TRIAL: NCT01956877
Title: Assessment of Normal Values of Esophagogastric Junction (EGJ) Distensibility in Healthy Volunteers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL45176.068.13
Record Dates: First submitted 2013-09-16; First posted 2013-10-08 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Healthy volunteers

SUMMARY:
To assess normal values of EGJ distensibility in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. No history of gastrointestinal disease, especially gastro-esophageal reflux disease
2. BMI = 18-30 kg/m²
3. Caucasian race
4. Subject signed the informed consent form and is able to adhere to study protocol

Exclusion Criteria:

1. Age < 18 years
2. Previous esophageal or gastric surgery
3. Co-morbidities (including cardiopulmonary disease, collagen diseases, obesity, coagulation disorders and co-morbidity hindering upper gastrointestinal endoscopy)
4. Patients using anticoagulants
5. Patients unable to give informed consent
6. Smoking
7. History of alcohol abuse or current excessive alcohol consumption (> 2 alcoholic beverages per day or > 14 alcoholic beverages per week)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 15 healthy volunteers, age > years
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
normal values of esophagogastric junction (EGJ) distensibility (mm2/mmHg) in healthy volunteers as measured with the EndoFLIP device | 3 months
  EGJ distensibility as measured by the index of the narrowest cross sectional area (mm2) and the corresponding intrabag pressure (mmHg)

SECONDARY OUTCOMES:
Establishing a cut-off value of EGJ distensibility (mm2/mmHg) based on the 90% percentile distribution of measurements performed in healthy volunteers. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands